CLINICAL TRIAL: NCT02817334
Title: A Prospective Clinical Study for Evaluation of Safe Resection Margin in Breast Conserving Surgery
Brief Title: A Prospective Clinical Study for Evaluation of Safe Resection Margin in Breast Conserving Surgery in Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, So-Youn Jung, Medical Doctor, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC-1410202-3
Record Dates: First submitted 2016-06-01; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
Keywords: Near-infrared fluorescence; Indocyanine green, ICG; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- indocyanine green (Experimental): As inject only indocyanine green (ICG), it provide the surgeon visual guidance to ensure better outcome.
  Intervention: Drug: indocyanine green
  Interventions: Drug: indocyanine green

INTERVENTIONS:
Drug: indocyanine green — As inject only indocyanine green (ICG), it provide the surgeon visual guidance to ensure better outcome.
  Other Names: Near-infrared fluorescence

SUMMARY:
Near-infrared (NIR) fluorescence imaging using indocyanine green (ICG) has been used for breast cancer surgery such as sentinel lymph node (SLN) mapping and breast cancer localization.

In this study, our hypothesis are as following:

1. As inject only indocyanine green (ICG), it provide the surgeon visual guidance to ensure better outcome.
2. indocyanine green (ICG) permitted accurate preoperative and intraoperative detection of the SLNs as well as nonpalpable benign brest lesion in patients with breast cancer.

DETAILED DESCRIPTION:
Indocyanine green, ICG (ICG-fluorescence)

* ICG is the most commonly used fluorophore which approve by FDA.
* NIR-F imaging with ICG could be used in various surgeries. For example, SLN mapping in breast cancer and localization of liver metastasis, especially superficial lesion
* Contains sodium iodide, patients who have history of allergy to iodides should be used as caution.

Nonpalpable benign brest lesion localization

* New method for the localization and resection of non-palpable breast lesions.
* The breast lesion was correctly localized, and the area of ICG corresponded well to the site of the lesions.

ELIGIBILITY:
Inclusion Criteria:

* nonpalpable breast tumor < 5cm in patients with breast cancer.
* consented patients with more than 18 years
* Eastern Cooperative Oncology Group Performance status 0 or 1
* patients who need breast biopsy as treatment for breast cancer.

Exclusion Criteria:

* nonpalpable breast tumor ≥ 5cm in patients with breast cancer.
* inflammatory cancer of breast or patients who need MRM
* pregnancy
* history of severe allergy to ICG(Indocyanine Green)
* iode hypersensitiveness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
detection rate | one day
  after complete resection with intraoperative ultrasound confirmed the lesion

SECONDARY OUTCOMES:
determine the pathological stability | one day
  determine the pathological stability with biopsy results confirmed during surgery

OTHER OUTCOMES:
Side effects and availability Side effects and availability Side effects and availability side effects and availability | following up a week to 3 month
  Itchiness, erythema, rash and other allergic reactions there could have shots later.
  Itchiness, erythema, rash and other allergic reactions there could have shots later.
  Itchiness, erythema, rash and other allergic reactions there could have shots later.
  Itchiness, erythema, rash and other allergic reactions there could have shots later.
side effects and availability | following up a week to 3 month
  After scanning, difficulty breathing, a decrease in blood pressure checked whether he had o reaction, such as anaphylactic shock.
side effects ans availability | following up a week to 3 month
  The skin discoloration, verify that there aren't stay in a follow-up after three months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: So-Youn Jung, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea